CLINICAL TRIAL: NCT03232346
Title: A Strategy to Improve Success of Treatment Discontinuation in Buprenorphine Responders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7522; 1R21DA042243 (NIH)
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Opioid-use Disorder
Keywords: buprenorphine; naltrexone; Vivitrol; opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regimen 1 (Experimental): Rapid Monday to Friday oral naltrexone-induction procedure
  Interventions: Drug: Vivitrol
- Regimen 2 (Experimental): 5-week buprenorphine taper from maintenance dose of 8, 6, or 4mg
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Vivitrol — Oral naltrexone induction procedure followed by Vivitrol
  Arms: Regimen 1
Drug: Buprenorphine — 5-week buprenorphine taper
  Arms: Regimen 2

SUMMARY:
This study is an open--label randomized outpatient trial to evaluate feasibility and efficacy of rapid buprenorphine (BUP) discontinuation followed by brief course of treatment with long--acting naltrexone (XR--NTX) and to compare it to the standard method of gradual BUP taper.Individuals with opioid use disorder (OUD) (N=60) who have successfully completed at least 6 months of buprenorphine treatment and do not wish to remain in a long--term buprenorphine maintenance program will be recruited. The first phase includes a 4--week period of stabilization on buprenorphine 4--8 mg at the research clinic to assure that patients are stable, compliant, and free from illicit opioids. Participants that meet the above criteria will be randomized 1:1 to: 1) buprenorphine discontinuation and outpatient transition to XR--NTX with 3 monthly injections, or 2) buprenorphine discontinuation using a gradual 5-week long taper. In both groups participants will receive weekly relapse prevention therapy and will be monitored for the duration of the trial, which is 25 weeks post randomization.

ELIGIBILITY:
Inclusion Criteria:

1. A documented history of treatment with buprenorphine or buprenorphine/naloxone for at least 6 months with sustained abstinence from illicit opioids for at least 3 months. Participants must be maintained on daily dose of buprenorphine in the 4--8 mg range.(MINI interview by therapist, Clinical interview by psychiatrist, consultation with previous prescriber or the verification patients's self-report with the prescribing records (PMP) with patient's permission).
2. Aged 18 to 60 years (Clinical interview).
3. In otherwise good health based on complete medical history, physical examination, vital signs measurement, ECG, and laboratory tests (hematology, blood chemistry, urinalysis) within normal ranges (Medical history and physical examination by psychiatrist or NP, laboratory tests (serum Chem-20 and CBC, urinalysis), ECG).
4. Seeking buprenorphine discontinuation and willing to accept randomization to either taper from buprenorphine or injection naltrexone (clinical interview).

Exclusion Criteria:

1. Lifetime history of DSM-5 diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder (MINI interview by therapist, Clinical interview by psychiatrist).
2. Current DSM-5 criteria for any other psychiatric disorder that in the investigator's judgment is unstable, would be disrupted by the study medication, or is likely to require pharmacotherapy or psychotherapy during the study period. Concurrent treatment with other psychotropic medication is exclusionary. ( MINI interview by therapist, Clinical interview and mental status exam by psychiatrist, contact with collateral information as needed and available).
3. Individuals who meet DSM-5 criteria for any substance use disorders - severe, other than opioid and nicotine use disorder. Physiological dependence on alcohol or sedative-hypnotics is exclusionary. (MINI interview by therapist, Clinical interview by psychiatrist).
4. A recent history of binge-use of alcohol or sedative-hypnotics (using large amounts in a short time to severe intoxication or blackouts). (Clinical interview by psychiatrist).
5. Pregnancy, lactation, or failure to use adequate contraceptive method in female patients who are currently engaging in sexual activity with men. ( Clinical interview by psychiatrist, physical examination and medical history by psychiatrist or NP, urine pregnancy test, serum HCG).
6. Unstable medical conditions, such as AIDS, cancer, uncontrolled hypertension (blood pressure > 140/90), uncontrolled diabetes, pulmonary hypertension or heart disease. (Medical history and physical examination by psychiatrist or NP, laboratory tests (serum Chem-20 and CBC, urinalysis), ECG).
7. Legally mandated to participate in a substance use disorder treatment program ( Participant self-report, Clinical interview by psychiatrist).
8. Current or recent history of significant violent or suicidal behavior, risk for suicide or homicide (MINI interview by therapist, Clinical interview by psychiatrist).
9. History of accidental opioid overdose in the last three years or any other significant history of overdose following detoxification within past 10 years defined as an episode of opioid-induced unconsciousness, whether or not medical treatment was sought or received. ( MINI interview by therapist, Clinical interview by psychiatrist).
10. Elevated liver function tests (AST and ALT > 3 times the upper limit of normal) ( Laboratory tests -serum Chem-20).
11. Known history of allergy, intolerance, or hypersensitivity to naltrexone or any other study medications( Participant self-report, Clinical interview by psychiatrist).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen 1 | Regimen 2
Started | 6 | 5
Completed | 2 | 3
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 | Regimen 2 | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 41.7 [29 to 52] | 49.6 [35 to 60] | 45.3 [29 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Successfully Transitioned Off Buprenorphine
Description: Percent of patients retained in treatment and abstinent from opioids at the end of the trial
Time Frame: Week 25
Population: Participants who were randomized to one of the two study regimens
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 | Regimen 2
Number analyzed (Participants) | 6 | 5
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Regimen 1 | Regimen 2
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen 1 (N=6) | Regimen 2 (N=5)
hospitalization for pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant had difficulty breathing, chest congestion, runny nose, and decreased energy. The participant was admitted to the hospital, and he was diagnosed with pneumonia. Participant was treated with IV antibiotics and fully recovered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03232346/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03232346/SAP_001.pdf